CLINICAL TRIAL: NCT03834571
Title: A Randomized Phase II Trial of Concurrent Chemotherapy and Pelvic Radiation Therapy With or Without Paclitaxel and Carboplatin in HIV-positive Women With Locally Advanced Cervical Cancer (LACC)
Brief Title: Testing the Addition of Paclitaxel and Carboplatin Given After Standard Chemotherapy and Radiation for Cervical Cancer in HIV-positive Women
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Not approved by CTEP
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry); University of Stellenbosch (Other); University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC-102; NCI-2018-01903 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AMC-102 (Other: AIDS Malignancy Consortium); AMC-102 (Other: CTEP); UM1CA121947 (NIH)
Record Dates: First submitted 2019-02-06; First posted 2019-02-08 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Squamous Cell Carcinoma, Not Otherwise Specified; FIGO Stage IIB Cervix Carcinoma; FIGO Stage III Cervix Carcinoma; FIGO Stage IVA Cervix Carcinoma; HIV Infection
Keywords: Cervical Cancer; HIV Infection
MeSH Terms: conditions — HIV Infections; Uterine Cervical Neoplasms | interventions — Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Paclitaxel; Taxes; Remote Patient Monitoring; Radiotherapy; Radiation

STUDY DESIGN:
Intervention Model Description: All participants will receive standard chemotherapy and radiation for the first 8 weeks of the trial. Four (4) to 8 weeks after finishing standard therapy, participants meeting eligibility criteria for randomization will be assigned to 1 of 2 arms. Arm 1 will receive up to 4 cycles of adjuvant IV chemotherapy (carboplatin and paclitaxel, 21-day cycle length), and arm 2 will undergo active monitoring for cancer recurrence or progression. All participants will be monitored every 3 months for recurrence or progression through 2 years after study enrollment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I (standard care, carboplatin, paclitaxel) (Experimental): STANDARD CARE: Patients receive cisplatin IV over 30-60 minutes on days 1, 8, 15, 22, 29, and 36. Patients also undergo radiation therapy over 2-5 fractions 5 days a week for up to 8 weeks in the absence if disease progression or unacceptable toxicity. 4-8 weeks following standard of care.
  4-8 weeks following standard care, patients receive carboplatin IV over 1 hour and paclitaxel IV over 3 hours on day 1. Courses repeat every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Paclitaxel; Radiation: Radiation Therapy
- Arm II (standard care, active monitoring) (Active Comparator): STANDARD CARE: Patients receive cisplatin IV over 30-60 minutes on days 1, 8, 15, 22, 29, and 36. Patients also undergo radiation therapy over 2-5 fractions 5 days a week for up to 8 weeks in the absence if disease progression or unacceptable toxicity. 4-8 weeks following standard of care.
  4-8 weeks following standard care, patients undergo active monitoring at 3, 6, 9, 12, 18 and 24 months.
  Interventions: Drug: Cisplatin; Procedure: Patient Monitoring; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm I (standard care, carboplatin, paclitaxel)
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm I (standard care, carboplatin, paclitaxel)
Procedure: Patient Monitoring — Undergo active monitoring
  Other Names: monitor
  Arms: Arm II (standard care, active monitoring)
Radiation: Radiation Therapy — Undergo radiation
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; RADIOTHERAPY; RT; Therapy, Radiation

SUMMARY:
This phase II trial studies how well standard chemotherapy and radiation therapy given with or without paclitaxel and carboplatin work in treating human immunodeficiency virus (HIV)-positive women with cervical cancer that has spread to nearby tissue or lymph nodes. Drugs used in chemotherapy, such as cisplatin, paclitaxel, and carboplatin work in different ways to stop the growth of tumor cells. They may either kill the cancer cells by stopping them from dividing, or by stopping them from spreading. Radiation therapy to the pelvis destroys potential cancer cells in the pelvic area and significantly reduces the risk of tumor recurrence in the pelvic area. It is not yet known if giving chemotherapy and radiation therapy with paclitaxel and carboplatin afterward may work better than than just chemotherapy and radiation therapy in treating HIV-positive patients with advanced cervical cancer.

DETAILED DESCRIPTION:
STANDARD CARE: All participants receive cisplatin intravenously (IV) over 30-60 minutes on days 1, 8, 15, 22, 29, and 36. Patients also undergo radiation therapy over 2-5 fractions for 5 days a week, for up to 8 weeks in the absence of disease progression or unacceptable toxicity. Four (4) to 8 weeks after finishing standard chemotherapy and radiation, participants are randomized to 1 of 2 arms.

RANDOMIZED ARMS:

Arm I: Patients receive carboplatin IV over 1 hour and paclitaxel IV over 3 hours on day 1. Courses repeat every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Participants are followed at 3, 6, 9, 12, 18 and 24 months for recurrence or progression.

Arm II: Participants undergo active monitoring at 3, 6, 9, 12, 18 and 24 months for recurrence or progression.

ELIGIBILITY:
This trial will be conducted at selected AIDS Malignancy Consortium sites in Sub-Saharan Africa.

Eligibility Criteria for Screening

* Ability to understand and the willingness to provide informed consent.
* Participant has clinically diagnosed LACC and self-reports as HIV-positive
* Age ≥ 18 years. DOB and age will be determined based on best possible information or documentation available.
* ECOG performance status ≤ 2 (Karnofsky ≥ 50%, see Appendix III).

Inclusion Criteria for chemoradiation treatment enrollment:

* Participants with locally advanced primary, untreated, histologically-confirmed, documented invasive squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma of the uterine cervix, adequately clinically staged by standard clinical guidelines, with Federation of Gynecology and Obstetrics (FIGO) stages IIB, III, or IVA
* HIV positive. Documentation of HIV-1 infection by means of any one of the following:

  * Documentation of receipt of ART by a licensed health care provider (documentation may be a record of an ART prescription in the participant's medical record, a written prescription in the name of the participant for ART, or pill bottles for ART with a label showing the participant's name)
  * HIV-1 ribonucleic acid (RNA) detection by a licensed HIV-1 RNA assay demonstrating >1000 RNA copies/mL confirmed by a licensed screening antibody and/or HIV antibody antigen combination assay
  * Any licensed HIV screening antibody and/or HIV antibody/antigen combination assay confirmed by a second licensed HIV assay such as a HIV-1 Western blot confirmation or HIV rapid multispot antibody differentiation assay.

    * Note: The term "licensed" refers to a kit that has been certified or licensed by an oversight body within the participating country and validated internally. WHO (World Health Organization) and CDC (Centers for Disease Control and Prevention) guidelines mandate that confirmation of the initial test result must use a test that is different from the one used for the initial assessment. A reactive initial rapid test should be confirmed by either another type of rapid assay or an E/CIA that is based on a different antigen preparation and/or different test principle (e.g., indirect versus competitive), or a Western blot or a plasma HIV-1 RNA viral load.
* Hemoglobin >= 10 g/dL (6.2 mmol/L) (participants receiving transfusion are permitted) (within 4 weeks prior to enrollment)
* Leukocytes: >= 3,000/mm^3 (3.0 x 10^9/L) (within 4 weeks prior to enrollment)
* Absolute neutrophil count: >= 1,500/mm^3 (1.5 x 10^9/L) (within 4 weeks prior to enrollment)
* Platelets: >= 100,000/mm^3 (100 x 10^9/L) (within 4 weeks prior to enrollment)
* CD4 T-cell count a minimum of 200 cells/uL (within 4 weeks prior to enrollment)
* Total bilirubin =< 2 x institutional upper limit of normal (ULN) unless related to antiretroviral use (e.g., atazanavir or indinavir), then the direct bilirubin must be =< 2 x ULN (within 4 weeks prior to enrollment)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]): =< 3 x ULN (within 4 weeks prior to enrollment)
* Creatinine levels within normal institutional limits or, creatinine clearance >= 60 mL/min/1.73 m^2 (1.00 mL/s) calculated by the Cockcroft-Gault equation for women for participants with creatinine levels above institutional normal (within 4 weeks prior to enrollment)
* All participants must be prescribed combination antiretroviral therapy with the goal of virological suppression using an acceptable regimen that adheres to national guidelines for treatment of HIV infection. If on a ritonavir- or cobicistat-based regimen, the participant must be switched to a non-ritonavir/ cobicistat-based regimen at least 7 days before treatment enrollment. Participants not on ART must start an acceptable regimen at least 7 days before treatment enrollment.
* In the investigator's opinion the participant is suitable for treatment with radical intent using concurrent chemotherapy and pelvic radiation followed by adjuvant chemotherapy
* Participants of childbearing potential, defined as a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months), must have a negative urine or serum pregnancy test within 3 weeks prior to enrollment and agree to use an effective form of contraception (e.g., barrier contraception, highly effective hormonal contraception) for the duration of treatment and for 6 weeks after stopping treatment
* Life expectancy of greater than 6 months

Exclusion Criteria for chemoradiation treatment enrollment:

* Participants who have had chemotherapy for cervical cancer within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Participants who are receiving any other investigational agents
* Participants who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicity > grade 1).
* Participants who have undergone hysterectomy including supracervical hysterectomy
* Acute active (such as tuberculosis or malaria), serious, uncontrolled infection
* Prior invasive malignancy requiring systemic chemotherapy diagnosed within the past 24 months (other than LACC)
* A medical or psychiatric illness that precludes ability to give informed consent or is likely to interfere with the ability to comply with the protocol stipulations
* Participants with circumstances that will not permit completion of the study or required follow-up. For instance, if travel to and from treatment site is an issue
* Participants with carcinoma of the cervical stump
* Participants with history of cardiovascular disease manifested as:

  * History of myocardial infarction
  * Unstable angina
  * Currently taking medication for treatment of angina
  * History of coronary artery bypass surgery
  * New York Heart Association class 3 or 4 heart failure
* Participants with enlarged para-aortic lymph node involvement above L3 on imaging that are suspicious for metastasis
* History of allergic reactions attributed to compounds of similar chemical or biological composition to study drugs (cisplatin, carboplatin, and paclitaxel)
* Participants who are breastfeeding a child. Cisplatin is known to be excreted in human milk.

Eligibility for Randomization

* Participants must have organ and marrow function within the following parameters within 4-8 weeks post CDDP/RT to be eligible for randomization
* Absolute neutrophil count: ≥1,500/mm3 (1.5 x 109/L)
* Platelets: ≥ 100,000/mm3 (100 x 109/L)
* CD4 T-cell > 100 cells/µL
* HIV viral load < 400 copies/mL
* ECOG performance status ≤ 2 (Karnofsky ≥ 50%).
* Successful completion of CDDP/RT, defined as receiving 4-6 cycles of cisplatin and completion of the equivalent dose per fraction of >78 Gy to Point A.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-31 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) evaluated using Response Evaluation Criteria in Solid Tumors 1.1 | The time from registration enrollment to disease recurrence, disease progression, or death for any reason, assessed up to 2 years
  The intervention arm will be compared to the control arm for improvement in PFS via one-sided log-rank test. This test will be conducted once for the interim analysis and once for the final analysis.

SECONDARY OUTCOMES:
Incidence of adverse events graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | Up to 2 years
  The frequency of adverse events (AEs) and their severity will be tabulated to evaluate the safety and tolerability. Safety and tolerability will be evaluated through tracking the number of dose delays, dose reductions, missing doses, and number of doses received and compliance.
Progression free survival by stage | Up to 2 years
  The Kaplan Meier method will be used to estimate the 2-year PFS and corresponding 95% confidence intervals of human immunodeficiency virus (HIV)-infected women with locally advanced cervical cancer (LACC) treated on study, stratified by FIGO 2018 stage.
Treatment effect on participants HIV disease status by assessing CD4 counts | Up to 2 years
  Descriptive statistics will be used to describe the effects of treatment on participants' HIV disease status by assessing CD4 counts.
Treatment effect on HIV disease status by assessing HIV viral load | Up to 2 years
  Descriptive statistics will be used to describe the effects of treatment on participants' HIV disease status by assessing HIV viral load.
Cervical cancer recurrence patterns | Up to 2 years
  Binomial proportions and their corresponding 95% confidence intervals will be used to describe cervical cancer recurrence patterns in HIV-infected participants with LACC defined as loco-regional and/or distant recurrences.
Overall survival (OS) | From entry to protocol to death; or for living participants, the date of last contact, assessed up to 2 years
  The Kaplan Meier method and corresponding 95% confidence interval will be used to estimate the overall survival. The causes of death will be listed.
Progression free survival (PFS) in women not meeting criteria for randomization by stage | Up to 2 years
  The Kaplan Meier method will be used to estimate the 2-year PFS and corresponding 95% confidence intervals of HIV-infected women with LACC treated on study but who did not meet the eligibility criteria for randomization, stratified by FIGO 2018 stage.

OTHER OUTCOMES:
Evaluation of cervical human papilloma virus (HPV) types | Up to 2 years
  Counts and binomial proportions will be used to evaluate the cervical HPV types present in the HIV-positive women with cervical cancer.
Persistence of cervical HPV pre-treatment | Up to 2 years
  McNemar's test will be used to assess persistence of cervical HPV pre-treatment.
Persistence of cervical HPV post-treatment | Up to 2 years
  McNemar's test will be used to assess persistence of cervical HPV post-treatment.
Presence of HPV in the anus pre-treatment | Up to 2 years
  McNemar's test will be used to assess the presence of HPV in the anus pre-treatment.
Presence of HPV in the anus post-treatment | Up to 2 years
  McNemar's test will be used to assess the presence of HPV in the anus post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ntokozo Ndlovu, Principal Investigator — Parirenyatwa Hospital
Locations (3):
- South Africa (2):
  - Stellenbosch University, Cape Town
  - University of Witwatersrand, Johannesburg
- Parirenyatwa Hospital, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: No